CLINICAL TRIAL: NCT05571644
Title: Neoadjuvant Treatment With mFOLFOXIRI Plus Cadonilimab (AK104) Versus mFOLFOX6 Alone in Locally Advanced Colorectal Cancer: a Randomized Control Phase II Study (OPTICAL-2)
Brief Title: Neoadjuvant Treatment With mFOLFOXIRI Plus Cadonilimab (AK104) Versus mFOLFOX6 in Locally Advanced Colorectal Cancer
Acronym: OPTICAL-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-15
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: Neoadjuvant therapy; mFOLFOXIRI; Cadonilimab (AK104); mFOLFOX6
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- mFOLFOXIRI+Cadonilimab (Experimental): Patients will receive neoadjuvant treatment with mFOLFOXIRI plus cadonilimab for 6 cycles before surgey
  Interventions: Drug: mFOLFOXIRI + Cadonilimab
- mFOLFOX6 (Active Comparator): Patients will receive neoadjuvant mFOLFOX6 chemotherapy every two weeks for 6 cycles before surgery.
  Interventions: Drug: mFOLFOX6
- mFOLFOXIRI (Active Comparator): Patients will receive neoadjuvant mFOLFOXIRI chemotherapy every two weeks for 6 cycles before surgery.
  Interventions: Drug: mFOLFOXIRI
- mFOLFOXIRI+AK104+fruquintinib (Other): Therapeutic Exploratory：Patients will receive neoadjuvant treatment with mFOLFOXIRI plus cadonilimab for 6 cycles and fruquintinib (3mg Qd, D1-21, Q4W for 3 months) before surgey
  Interventions: Drug: mFOLFOXIRI+AK104+fruquintinib

INTERVENTIONS:
Drug: mFOLFOXIRI + Cadonilimab — Cadonilimab（AK104）6mg/kg, intravenous d for 60 minutes, followed by mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) every 2 weeks for 6 cycles before surgery
  Other Names: Oxaliplatin; Irinotecan; 5-Fluorouracil; Leucovorin; Cadonilimab (AK104)
  Arms: mFOLFOXIRI+Cadonilimab
Drug: mFOLFOX6 — mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) every 2 weeks for 6 cycels before surgery
  Other Names: Oxaliplatin; 5-Fluorouracil; Leucovorin
  Arms: mFOLFOX6
Drug: mFOLFOXIRI — mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) every 2 weeks for 6 cycles before surgery
  Other Names: Oxaliplatin; Irinotecan; 5-Fluorouracil
  Arms: mFOLFOXIRI
Drug: mFOLFOXIRI+AK104+fruquintinib — Cadonilimab（AK104）6mg/kg, intravenous d for 60 minutes, followed by mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) every 2 weeks for 6 cycles, and fruquintinib (3mg Qd, D1-21, Q4W for 3 months) before surgery
  Arms: mFOLFOXIRI+AK104+fruquintinib

SUMMARY:
Neoadjuvant chemoradiotherapy (CRT) followed by total mesenteric excision (TME) and adjuvant chemotherapy was the standard of treatment for locally advanced rectal cancer (LARC) in the past two decades. The main obstacles for improving survival benefit of LARC was distant metastasis. Recently, total neoadjuvant therapy (TNT) had been recommended as new preferred option for LARC. Induction chemotherapy with FOLFOXIRI followed by CRT or short-course radiotherapy followed by FOLFOX chemotherapy had improved survival benefit for LARC.

Neoadjuvant immunotherapy had also been explored in pMMR patients with CRC. In the NICHE trial, neoadjuvant therapy with 2 dose of nivolumab and 1 dose of ipilimumab led to 29% of pathological response and 13% of pCR. Cadonilimab (AK104) was a PD-1/CTLA-4 bi-specific antibody. Here, we tried to explore the efficacy of Neoadjuvant Treatment With mFOLFOXIRI with or without Cadonilimab (AK104) Versus mFOLFOX6 in LARC.

DETAILED DESCRIPTION:
This study was a prospective, randomized, uncontrolled phase II trial to evaluate the efficacy of mFOLFOXIRI combined with AK104 neoadjuvant therapy versus mFOLFOX6 neoadjuvant therapy in LARC.

The inclusion criteria: locally advanced colon cancer (T3>5mm or T4 on enhanced CT assessment, with distant metastasis excluded); Locally advanced rectal cancer (pelvic MR assessment as stage ii-iii, less than 12cm from the anal margin, no distant metastasis).

Group A: mFOLFOXIRI combined with Cadonilimab (AK104) for 6 cycles before surgery

Group B: 6 cycles of neoadjuvant chemotherapy with mFOLFOX6 before surgery

Group C: 6 cycles of neoadjuvant chemotherapy with mFOLFOXIRI before surgery

Group D (exploratory cohort): mFOLFOXIRI combined with Cadonilimab (AK104) and fruquintinib for 3 months before surgery (not for randomised)

All groups were re-evaluated after 3 cycles and 6 cycles of treatment. If surgery was feasible after multidisciplinary evaluation, TME resection was performed, and adjuvant treatment was performed according to standard treatment after operation. For locally advanced rectal cancer, preoperative pelvic enhanced MRI was used to evaluate tumor regression after 6 cycles of preoperative treatment. For patients who still had MRF+ and/or T4 after treatment, additional short-course radiotherapy was allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70;
2. Colorectal adenocarcinoma with definite histological evidence;
3. ECOG Performance status score is 0-1
4. Colon cancer was evaluated as T3>5mm or T4 by contrast-enhanced CT examination of the chest, abdomen and pelvis, and distant displacement was excluded; Rectal cancer was graded as T3-4 and/or N+ by pelvic contrast-enhanced MRI examination, and the lower margin of the tumor was less than 12cm away from the anal margin. Distant metastasis was excluded by chest, abdomen and pelvis CT.
5. The primary rectal tumor was assessed as complete resections by a multidisciplinary collaboration group on colorectal cancer, including at least 2 gastrointestinal surgeons and 1 radiologist;
6. No previous systemic antitumor therapy for colorectal cancer, including cytotoxic drugs, immunotherapy, molecular targeted therapy, etc.;
7. Adequate organ function based on the following laboratory test values obtained within 7 days prior to treatment:

   Hemoglobin ≥90g/L, neutrophil count ≥1.5×109/L, platelet count ≥75×109/L, serum total bilirubin ≤1.5× upper limit of normal value (UNL), aspartate transferase ≤2×UNL, alanine transferase ≤3×UNL, serum creatinine ≤1.5×UNL;
8. Willing and able to comply with research protocols and visit plans.

Exclusion Criteria:

1. The patient was complicated with obstruction, active bleeding, or perforation and required emergency surgery or stent placement;
2. Active, known or suspected autoimmune diseases (except type I diabetes, residual hypothyroidism requiring only hormone replacement due to autoimmune conditions, or autoimmune diseases that are not expected to recur in the absence of external triggers);
3. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C, defined as HCV-RNA above the detection limit of the assay) or co-infection with hepatitis B and C;
4. Known allergy to the treatment drug or allergy or intolerance to its ingredients;
5. Major surgery or severe trauma, such as laparotomy, thoracotomy, laparoscopic organ resection, etc. within the previous 4 weeks (the surgical incision should be completely healed before enrollment);
6. Existing or coexisting other active malignancies (except those that have been treated with curative therapy and remain disease-free for more than 5 years or carcinoma in situ that can be cured by adequate treatment);
7. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody and anti-cytotoxic T-lymphocyte-associated protein 4 (Cytotoxic T-lymphocyte-associated protein 4) antibody. Ctla-4) antibodies or other drugs/antibodies that act on T-cell costimulatory or checkpoint pathways;
8. Had active coronary artery disease, severe/unstable angina pectoris or newly diagnosed angina pectoris or myocardial infarction within 6 months prior to study enrollment; Thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis, occurred within the previous 6 months;
9. The New York Heart Association (NYHA) class II or higher congestive Heart failure (see Appendix 3);
10. Presence of active inflammatory bowel disease or other colorectal disease leading to chronic diarrhea;
11. The presence of any toxicity (Common Terminology Criteria for Adverse Events, CTCAE) (version 5.0) grade 1 or above (except anemia, alopecia, and skin pigmentation) caused by previous treatment that has not subsided;
12. Previous or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of pulmonary function and other lung diseases;
13. Active tuberculosis (TB), receiving anti-TB therapy or receiving anti-TB therapy within 1 year before the first dose;
14. Persons with known syphilis infection requiring treatment;
15. Had used immunosuppressive drugs within 4 weeks before the first dose, Does not include the nasal spray, inhalation, or other ways of topical corticosteroids or physiological doses of systemic corticosteroids (i.e., no more than 10 mg/day prednisone or other equivalent dose glucocorticoids), allows for prevention of allergic reactions, or treatment of diseases such as asthma, chronic obstructive pulmonary disease of breathing difficulties for the temporary use of glucocorticoid;
16. Receive live attenuated vaccine within 4 weeks before the first dose or during the study period;
17. Pregnant or lactating women; Women of reproductive age (< 2 years after last menstruation) who do not use or refuse to use effective non-hormonal contraception or men at risk of having children.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | 1 year
  Proportion of patients experiencing a pCR to preoperative treatment in each group

SECONDARY OUTCOMES:
Major pathological response rates | 1 year
  The proportion of patients experiencing a major pathological response (≤10% of residual viable tumor in the surgical specimen) to preopeartive treatment in each group
Disease-free survival (DFS) | 3 years
  Defined as the time from randomization to relapse, metastasis or death from any cause.
Local recurrence rate | 3 years
  Defined as the time from randomization to local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided